CLINICAL TRIAL: NCT06095414
Title: Prospective Study of MRI-based Radiomics in Breast Cancer
Brief Title: Prospective Radiomics Study for Breast Cancer
Status: Completed | Type: Observational
Sponsor: Korea University Ansan Hospital (Other)
Responsible Party: Principal Investigator, Bo Kyoung Seo, Professor, Korea University Ansan Hospital
Other Study IDs: KURADIOMICS
Record Dates: First submitted 2023-10-11; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MRI — MRI based assessment of tumor microenvironment in breast cancer mass

SUMMARY:
The goal of this prospective study is to develop MRI-based models representing tumor microenvironment in participants with invasive breast cancer.

The main purpose of this study is to analyze the association of diffusion-, T2-, and dynamic contrast-enhanced T1-weighted images of 3T MRI before treatment with the immunohistochemical reactivity of tumor microenvironment including the extracellular matrix and immune cells of core-needle biopsy specimens For this purpose, investigators extract 16145 radiomic features from the intratumoral and peritumoral regions on MRI of participants with invasive breast cancer before treatment.

DETAILED DESCRIPTION:
The written informed consents for the participation into this prospective study is done in participants who are diagnosed with invasive breast cancer before surgery with curative intent. After enrollment, breast MRI is done for particpants and diffusion-, T2-, and dynamic contrast-enhanced T1-weighted images are extracted from the results of MRI of participants. The tumor tissue samples are archived from participants before surgery through core-needle biopsy and the immunohistochemistry is done to assess the components of tumor microenvironment including intraturmoal and peritumoral components through volume histochemical assessment. Radiomic feature selection and prediction model building are performed using the least absolute shrinkage and selection operator and linear regression analysis, respectively. The investigators apply fivefold cross-validation to prevent overfitting, and the performance is evaluated using the area under the receiver operating characteristic curve (AUC) and the DeLong test.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with invaseiv breast cancer

Exclusion Criteria:

* Diagnosed with other cancers

Ages: 20 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population should fulfill the following criteria as follows:(a) histologically confirmed invasive breast cancer, (b) participant consent, and (c) MRI performed before treatment
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
The signal intensity of Magnetic Resonance Images for tumor microenvironment | Baseline, pre-surgery
  The percentage of diffusion-, T2-, and dynamic contrast-enhanced T1-weighted images correlated with the percentage of immune cells infiltrating tumor microenvironment of breast tumor tissue

CONTACTS AND LOCATIONS:
Overall Officials: Bo Kyoung Seo, MD., PhD, Principal Investigator — Korea University Ansan Hospital
Locations (1):
- Bo Kyoung Seo, Ansan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim ES, Ham S, Seo BK, Lee JY, Sun W, Jeon M, Joo M, Park S, Wang S, Lee B, Lee HY, Bae MS, Cho KR, Woo OH, Song SE, Kim SY. Optimized prediction of breast cancer tumor microenvironment using MRI-based intratumoral and peritumoral radiomics: a prospective study. Front Oncol. 2025 Nov 6;15:1654508. doi: 10.3389/fonc.2025.1654508. eCollection 2025. PMID 41278298